CLINICAL TRIAL: NCT05311605
Title: REperfusion Therapy for Acute Ischemic STrOke Due to Large aRtEry Occlusion
Acronym: RESTORE
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Beijing Municipal Science & Technology Commission (Other); Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Principal Investigator, Yunyun Xiong, Professor of Neurology and Stroke Center, Beijing Tiantan Hospital
Other Study IDs: KY-2022-029-01
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Vascular Occlusion; Endovascular Treatment; Mechanical Thrombectomy; Perfusion Imaging
Keywords: ischemic stroke; vascular occlusion; endovascular treatment; mechanical thrombectomy; perfusion imaging
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — serum sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to establish a clinical and advanced imaging database of acute ischemic stroke patients treated with mechanical thrombectomy due to large vessel occlusion of anterior circulation within 24 hours from stroke onset in China, and to investigate the predictors and potential mechanisms of futile recanalization after mechanical thrombectomy.

DETAILED DESCRIPTION:
The time-window of mechanical thrombectomy for ischemic stroke has extended from 4.5 hours to 24 hours based on the results of the DAWN and DEFUSE 3 trials. However, evidence on the effectiveness and safety of mechanical thrombectomy within 24 hours in the real-world is insufficient.

This is a multi-center, prospective, registry cohort study that acute ischemic stroke patients treated with mechanical thrombectomy due to large vessel occlusion of anterior circulation within 24 hours from stroke onset in China. A retrospective dataset was also build in these stroke centers for analysis. A total of 1600 patients with advanced imaging data were anticipated to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years;
* Perfusion imaging completed including CTA+CTP or MRA+PWI+DWI before thrombectomy
* Large vessel occlusion of cerebral anterior circulation (ICA, MCA-M1 or MCA-M2) confirmed by CTA or MRA, planned to receive or received stenting or aspiration thrombectomy
* Time intervals ≤ 24 hours from stroke onset to groin puncture.(fulfilled the inclusion of DAWN or DEFUSE 3 trial if the time intervals from stroke onset to groin puncture was ≥6 hours)
* mRS score ≤2 before admission
* Informed consent obtained for longitudinal enrolled patients, waived of consent for retrospectively included cases

Exclusion Criteria:

* Had a history of infective disease, immunity disease, radiotherapy at head or neck, carotid dissection or other carotid disease.
* Unable to receive CT or MR scan due to heart failure, cardiac pacemaker, metal implants or claustrophobia, etc.
* Unable to be injected with contrast agent due to allergy, renal dysfunction, etc.
* Unlikely to adhere to the study protocol or follow-up ( life expectancy ≤ 3 months)
* Already participated in other drug trials

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ischemic stroke patients that received mechanical thrombectomy due to large vessel occlusion of anterior circulation within 24 hours from stroke onset and had perfusion imaging both before and after thrombectomy.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Favorable functional outcome | 3 months from stroke onset
  proportion of mRS score 0-2 at 3 months. The modified Rankin Scale (mRS) has a minimum value of 0 and maximum value of 6. Higher value indicated worse functional outcome

SECONDARY OUTCOMES:
Excellent functional outcome at 90 days | 3 months from stroke onset
  proportion of mRS score 0-1 at 3 months
Ordinal distribution of mRS at 90 days | 3 months from stroke onset
  Number of participants with the ordinal distribution of mRS at 90 days
EQ-5D score at at 90 days | 3 months from stroke onset
  EQ-5D score at 3 months. EuroQol Five Dimensions Questionnaire scale (EQ-5D score) has a minimum value of 0 and maximum value of 100. Lower value indicated worse functional outcome
Neurological improvement at 24 hours | 24 hours from stroke onset
  NIHSS score <=1 or improvement of NIHSS score>=4 compared with baseline NIHSS. National Institution Health Stroke Scale (NIHSS) has a minimum value of 0 and maximum value of 45. Higher value indicated worse severity of neurological impairment.
recanalization post-operation | (Day 0) immediately the surgeon thought the thrombectomy completed and performed a second cerebral angiography .
  proportion of eTICI 2b50/2c/3. Thrombectomy is a surgical operation using a retrieve stent or aspiration catheter to remove the thrombus inside an occluded vessel and achieve recanalization.The eTICI is a scale to assess the degree of recanalization. So, once the surgeon thought he completed the thrombectomy, he needed to perform a cerebral angiography to assess the degree of recanalization using eTICI.
recanalization at 24 hours | 24 hours after thrombectomy completed
  proportion of eTICI 2b50/2c/3

OTHER OUTCOMES:
Infarction volume at 24 hours | 24 hours after thrombectomy completed
  infarction volume: volume of the tissue with CBF <30% or ADC<600×10-6mm2/s
symptomatic intracerebral hemorrhage at 36 hours | 36 hours after thrombectomy completed
  symptomatic intracerebral hemorrhage based on Heidelberg criterion
Mortality at 90 days | 90 days after thrombectomy completed
  Mortality of all-cause

CONTACTS AND LOCATIONS:
Overall Officials: Yunyun Xiong, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Yunyun Xiong, Beijing, China